CLINICAL TRIAL: NCT05941338
Title: Prospective, One-arm, Phase II Clinical Study of Tirelizumab in Combination With Carboplatin and Albumin-binding Paclitaxel for Neoadjuvant Therapy in Patients With Resectable Squamous Cell Carcinoma of the Head and Neck
Brief Title: Tirelizumab in Combination With Carboplatin and Albumin-binding Paclitaxel for Neoadjuvant Therapy in HNSCC
Acronym: HNC-SYSU-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-159-01
Record Dates: First submitted 2023-06-05; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Oral Cancer
Keywords: head and neck squamous cell carcinoma; oral cancer; pd-1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Drug:Tirelizumab , Carboplatin,albumin-bound paclitaxel Patients receive Tirelizumab IV on day 1, albumin-bound paclitaxel IV on day 1 and carboplatin IV on day 1 . Treatment repeats every 21 days for up to 2cycles in the absence of disease progression or unacceptable toxicity. Then surgery.
  Interventions: Drug: Tirelizumab ,+Carboplatin+albumin-bound paclitaxel

INTERVENTIONS:
Drug: Tirelizumab ,+Carboplatin+albumin-bound paclitaxel — Sintilimab (IV), dose= 200mg , day=1 , cycle length: 21 days. Carboplatin (IV), dose=300mg/m2, day= 1, cycle length: 21 days. albumin-bound paclitaxel (IV), dose=260mg/m2, day= 1, cycle length: 21 days. Intervention: Drug: Sintilimab , Carboplatin, albumin-bound paclitaxel

SUMMARY:
In this study, 100 patients with resectable head and neck squamous cell carcinoma (oral squamous cell carcinoma and oropharyngeal squamous cell carcinoma) were enrolled, who were combined with tirelizumab, carboplatin and albumin-binding paclitaxel before and after surgery. Tumor tissues and paracancer tissues of patients were collected to observe the imaging and pathological changes before and after treatment. At the same time, clinical information of patients, such as pathological grade, stage, treatment, prognosis, serology, imaging, etc. were collected to evaluate the safety and feasibility of tirelizumab combined with carboplatin and albumin-binding paclitaxel for neoadjuvant therapy of resectable oral and oropharyngeal squamous cell carcinoma. This is a prospective, one-arm, phase II clinical study.

Purpose Main purpose The efficacy of Tirelizumab combined with carboplatin and albumin-paclitaxel in neoadjuvant therapy for resectable head and neck squamous cell carcinoma was evaluated by calculating the major pathological response (MPR) rates in the experimental group.

The severity of adverse events associated with neoadjuvant therapy will be graded according to NCI CTCAE (version 5.0) during the course of this study and during follow-up, the incidence of adverse events in the experimental and control groups will be compared, and the safety of neoadjuvant therapy with Tirelizumab combined with carboplatin and albumin-paclitaxel in resectable head and neck squamous cell carcinoma will be evaluated.

Secondary Purpose

1. One-year event survival rate and event-free survival (EFS) of enrolled patients were evaluated (five years);
2. Pathological complete response rate (pCR) of enrolled patients was evaluated (5 years);
3. pTR of enrolled patients was evaluated;
4. Overall survival (OS) of enrolled patients was evaluated (5 years);
5. Radiological response of enrolled patients was assessed;
6. The rate of operation delay of enrolled patients was evaluated;

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age ≤65 years of age;
* Cytological or histological diagnosis of surgically resectable squamous cell carcinoma of the head and neck with the following stages:

T3-4a, N0-2, M0;

* According to the solid tumor efficacy evaluation criteria (RECIST version 1.1), there was at least one radiologically measurable lesion; First-line patients: have not previously received any systemic antitumor therapy for advanced/metastatic disease. Patients who had previously received platinum-containing adjuvant/neoadjuvant chemotherapy, or had received radical chemoradiotherapy for advanced disease, if the interval between disease progression or recurrence and the end of the last chemotherapy drug treatment was at least 6 months, were allowed to be enrolled in this study.
* ECOG score 0-1;
* Expected survival time > 3 months;
* Adequate organ function, subject shall meet the following laboratory indicators:

  1. The absolute value of neutrophil granulocyte (ANC) ≥1.5x109/L in the last 14 days without the use of granulocyte colony stimulating factor;
  2. Platelets ≥100×109/L without blood transfusion in the past 14 days;
  3. Hemoglobin &gt without blood transfusion or use of erythropoietin within the last 14 days; 9g/dL;
  4. Total bilirubin ≤1.5× upper limit of normal value (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
  7. Good coagulation function, defined as International Standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. Subjects whose baseline TSH is outside the normal range can be enrolled if total T3 (or FT3) and FT4 are within the normal range;
  9. The myocardial enzyme profile was within the normal range (if the researchers comprehensively judged that the simple laboratory abnormality was not clinically significant, it was also allowed to be included);
  10. For female subjects of childbearing age, a urine or serum pregnancy test should be tested negative within 3 days prior to receiving the first study drug administration (day 1 of Cycle 1). If the urine pregnancy test results cannot be confirmed negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
  11. If there is a risk of conception, all subjects (male or female) shall use contraception with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last study drug administration (or 180 days after the last chemotherapeutic drug administration).

Exclusion Criteria:

* Malignant diseases other than head and neck squamous cell carcinoma diagnosed within 5 years prior to initial administration (excluding basal cell carcinoma of the skin after radical treatment, squamous epithelial carcinoma of the skin, and/or carcinoma in situ after radical excision);
* Currently participating in an interventional clinical study, or receiving other investigational drugs or using investigational devices within 4 weeks prior to initial dosing;
* Previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs that target another stimulus or synergistic inhibition of T cell receptors (e.g., CTLA-4, OX-40, CD137);
* Systemic treatment with Chinese patent drugs or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) with indications of anti-head and neck squamous cell carcinoma within 2 weeks before the first administration;
* An active autoimmune immune disease requiring systemic treatment (e.g. with disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to initial administration. Alternative therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* Was receiving systemic glucocorticoid therapy (excluding nasal, inhalation, or other routes of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days prior to initial administration; Note: Physiological doses of glucocorticoids (≤10 mg/ day of prednisone or equivalent) are permitted;
* Clinically uncontrollable pleural effusion/abdominal effusion (patients with no need to drain effusion or no significant increase of effusion after 3 days of stopping drainage could be included in the group);
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Those who are known to be allergic to the active ingredients or excipients of the drug in this study, Pabolizumab, carboplatin and albumin-binding paclitaxel;
* Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss);
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positive coupled with a detected HBV-DNA copy number greater than the upper limit of normal in the laboratory of the study center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1) HBV viral load &lt before initial administration; At 1000 copies /ml (200 IU/ml), subjects should receive anti-HBV therapy to avoid viral reactivation throughout the study treatment period 2) For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required

* Active HCV infected subjects (HCV antibody positive and HCV-RNA level above the lower limit of detection);
* Received live vaccine within 30 days prior to initial administration (cycle 1, day 1); Note: Inactivated injectable virus vaccine against seasonal influenza is permitted for 30 days prior to initial administration; But live attenuated influenza vaccines administered intranasally are not allowed.
* Pregnant or lactating women;
* There is any serious or uncontrolled systemic disease, such as:

  1. The resting electrocardiogram (ECG) presents significant and severely uncontrollable abnormalities in rhythm, conduction or morphology, such as complete left bundle branch block, Ⅱ degree or above heart block, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina pectoris, congestive heart failure, and NYHA grade ≥ 2 chronic heart failure;
  3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before treatment;
  4. Poor blood pressure control (systolic > 140 mmHg, diastolic > 90 mmHg);
  5. A history of non-infectious pneumonia requiring glucocorticoid therapy or clinically active interstitial lung disease within 1 year prior to initial administration;
  6. Active pulmonary tuberculosis;
  7. There is an active or uncontrolled infection that requires systemic treatment;
  8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
  11. Urine routine indicated urine protein ≥++, and confirmed 24 hours urine protein quantity > 1.0 g;
  12. Patients with mental disorders and unable to cooperate with treatment; 17. Medical history or evidence of disease that may interfere with test results, prevent participants from participating fully in the study, abnormal values of treatment or laboratory tests, or other conditions that the investigator considers unsuitable for enrollment. The Investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 6 weeks
  Pathologic response rate to neoadjuvant treatment in resected tumor and lymph nodes. The rate of major pathologic response, defined as <10% residual viable tumor cells in the resection specimen will be compared to historic data with neoadjuvant chemotherapy.
Adverse events graded by CTCAE v5.0 | 90 days after surgery
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).

SECONDARY OUTCOMES:
Pathologic complete response | 6 weeks
  The absence(percentage) of invasive/in situ cancer and/or axillary lymph nodes
Event-free survival (EFS) | 1 years and 5 years
  In cancer, the length of time after primary treatment for a cancer ends that the patient remains free of certain complications or events that the treatment was intended to prevent or delay.
Overall survival（OS） | 5 years
  The time(years) from day 1 of study treatment until death from any cause.
Operation delay rate | 2months
  Rate of patients with an Unplanned Delay to Surgery defined as any change to scheduled surgery date considered to be at least possibly related to neoadjuvant treatment.
Radiographic Response | 6 weeks
  Radiographic response(rate) to treatment as defined by RECIST 1.1.

OTHER OUTCOMES:
Exploratory purpose | 5 years
  For inclusion, group treatment was performed according to the guidelines, and stratification factors affecting immunotherapy prognosis and treatment plan were explored according to stratification. The stratification factors taken into consideration are: P16 status, smoking history, TNM stage, tumor reduction (MPR condition), presence of risk factors (according to the guidelines, risk factors are presence of episopercular invasion, positive incisal margin, proximal incisal margin, pT3 or pT4, pN2 or pN3 lymph nodes located in the IV and V regions of the neck, Nerve invasion, vascular invasion, etc.) and postoperative radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sun memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided